CLINICAL TRIAL: NCT04433897
Title: Observing the Effect of Hormonal Replacement Therapy on Nocturia in Postmenopausal Women
Brief Title: Effect of Hormonal Replacement Therapy on Nocturia in Postmenopausal Women
Acronym: HARALD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC 2018/0315 (BC-02592)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Oral estrogen + IUD: Women who opt to be treated for their postmenopausal symptoms using Oral estrogen + IUD
  Interventions: Other: Questionnaire
- Oral estrogen + hysterectomy: Women who opt to be treated for their postmenopausal symptoms using Oral estrogen + hysterectomy.
  Interventions: Other: Questionnaire
- Oral estrogen + oral progesterone: Women who opt to be treated for their postmenopausal symptoms using Oral estrogen + oral progesterone.
  Interventions: Other: Questionnaire
- Transdermal estrogen + IUD: Women who opt to be treated for their postmenopausal symptoms using transdermal estrogen + IUD.
  Interventions: Other: Questionnaire
- Transdermal estrogen + hysterectomy: Women who opt to be treated for their postmenopausal symptoms using transdermal estrogen + hysterectomy.
  Interventions: Other: Questionnaire
- Transdermal estrogen + oral progesteron: Women who opt to be treated for their postmenopausal symptoms using transdermal estrogen + oral progesteron
  Interventions: Other: Questionnaire
- SERM: Women who opt to be treated for their postmenopausal symptoms using SERM's
  Interventions: Other: Questionnaire
- Aromatase inhibitor: Women who opt to be treated for their postmenopausal symptoms using aromatase inhibitor.
  Interventions: Other: Questionnaire
- Duavive: Women who opt to be treated for their postmenopausal symptoms using duavive.
  Interventions: Other: Questionnaire
- No treatment: Women who opt not to be treated for their postmenopausal symptoms.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — All women fulfilled 3 questionairres
  * TANGO
  * ICIQ -N
  * Perceived Stress Scale

SUMMARY:
Aim of this study was to observe

The study was adjusted in two parts:

PART 1 is a crossectional study in which the prevalance, risk factors and etiology of nocturia among postmenopausal women is assessed.

PART 2 is a cohort study observing the impact of 10 different hormonal substitution therapies on nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal symptoms (hot flushes, atrophy, ..)
* All women were 'early' postmenopausal stages +1a,+1b or +1c as defined by the 'Stages of Reproductive Aging Workshop' (STRAW) criteria

Exclusion Criteria:

* Intake of HRT on the moment of inclusion
* women with thyroid dysfunction
* women using antihypertensive agents
* women with a history of psychiatric or neurological disorders
* women with a history of alcohol or drug addiction.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is specific for postmenopausal women
Study Population: Women who are biochochemically confirmed to be postmenopausal.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in nocturnal Frequency | 6 months after initiating therapy
  Change from baseline in nocturnal voiding episodes assessed via nycturia and menopause questionnaire

SECONDARY OUTCOMES:
Change in bother linked with nocturnal frequency | 6 months
  Change in VAS scale of bother linked with nocturnal frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided